CLINICAL TRIAL: NCT03708159
Title: Step-Down Neurostimulation to Maintain Response After Repetitive Transcranial Magnetic Stimulation (rTMS) Using Transcranial Direct Current Stimulation (tDCS): The START Study
Brief Title: Maintenance of Response After rTMS for Depression Using tDCS
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 063-2018
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
Keywords: tDCS; Mindfulness meditation; Home-based tDCS; rTMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Mindfulness; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active tDCS + mindfulness meditation (Experimental): Participants randomized to this group will receive active tDCS 3 times a week for approximately 3 months and then weekly for 3 months. After completing baseline procedures they will be trained how to apply the tDCS device themselves. The first 3-6 treatments will be completed at the hospital to ensure proper and safe application. Prior to taking the tDCS device home, they will pass the self-application scale adequately 3 times. Each treatment session lasts 30 minutes, during which, they will engage in mindfulness meditation.
  Interventions: Device: active tDCS + mindfulness meditation
- sham tDCS + mindfulness meditation (Sham Comparator): Participants randomized to this group will receive sham tDCS 3 times a week for approximately 3 months and then weekly for 3 months. After completing baseline procedures they will be trained how to apply the tDCS device themselves. The first 3-6 treatments will be completed at the hospital to ensure proper and safe application. Prior to taking the tDCS device home, they will pass the self-application scale adequately 3 times. Each treatment session lasts 30 minutes, during which, they will engage in mindfulness meditation.
  Interventions: Other: sham tDCS + mindfulness meditation

INTERVENTIONS:
Device: active tDCS + mindfulness meditation — Participants are provided with an activation code. This code will unlock a single session with the pre-set 30 minute duration and intensity (direct current 2mA, current density 0.80A/m2, with anode over the left and cathode over the right dorsolateral prefrontal cortex, respectively). These devices will be set to active. Each tDCS sessions will be delivered in combination with a guided mindfulness meditation that we have recorded.
  Other Names: Soterix tDCS mini-Clinical Trials system (mini-CT) - active
  Arms: active tDCS + mindfulness meditation
Other: sham tDCS + mindfulness meditation — Participants are provided with an activation code. This code will unlock a single session with the pre-set 30 minute duration and intensity (direct current 2mA, current density 0.80A/m2, with anode over the left and cathode over the right dorsolateral prefrontal cortex, respectively). These devices will be set to sham. Each tDCS sessions will be delivered in combination with a guided mindfulness meditation that we have recorded.
  Other Names: Soterix tDCS mini-Clinical Trials system (mini-CT) - sham
  Arms: sham tDCS + mindfulness meditation

SUMMARY:
This is a double-blind, multi-site, randomized controlled trial (RCT) that will recruit 200 participants.The purpose of the RCT will be to evaluate the efficacy of transcranial direct current stimulation (tDCS) in combination with mindfulness meditation compared to sham tDCS to maintain wellness following an acute course of repetitive transcranial magnetic stimulation (rTMS) for up to 6 months.

DETAILED DESCRIPTION:
Home-based tDCS (active vs. sham) will involve 30-min tDCS (3 days per week) for the first 3 months and once weekly for the subsequent 3 months, in combination with mindfulness mediation for the duration of tDCS each treatment. Subjects who miss 4 consecutive treatment days or 20 percent of total treatments will be exit the treatment intervention as it is our intention to encourage compliance with the proposed treatments to maintain optimal wellness.

Aim 1. To investigate the efficacy of at home maintenance tDCS for patients with MDD who have responded to a successful acute course of rTMS.

Hypothesis 1. Patients receiving tDCS will have a higher proportion of sustained responders or remitters after 6 months compared to sham tDCS.

Exploratory Aim 2. To investigate clinical predictors of sustained response to rTMS using tDCS Hypothesis 2. Remitters and those not on benzodiazepines will be associated with greater likelihood of sustained response.

ELIGIBILITY:
Inclusion Criteria:

1. History of Major Depressive Disorder with most recent depressive episode treated with acute rTMS
2. Individuals capable to provide consent who are receiving care as outpatients/research participants, and are now responders or remitters (defined by 50% improvement on any depression scale since the beginning of treatment and HRSD-17 ≤ 15, or an HRSD-17 score <8).
3. Age 18-85, inclusive.

Exclusion Criteria:

1. History of a DSM-IV substance use disorder within the past three months
2. Concomitant major unstable medical illness
3. DSM-IV diagnosis of any psychotic disorder, obsessive compulsive disorder, or post-traumatic stress disorder (current or within the last year) as confirmed by the Mini-International Neuropsychiatric Interview (MINI)
4. DSM-IV diagnosis of personality disorder as assessed by a study investigator
5. Any significant neurological disorder (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis)
6. Presenting with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, Cushing's disease)
7. Any intracranial implant (e.g., aneurysm clips, shunts, cochlear implants) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
8. Any dermatological disorder or any cuts/broken skin in the scalp region that may affect the safe delivery of the tDCS stimulus
9. Requiring a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of tDCS
10. The inability to communicate in spoken and written English fluently enough to complete the neuropsychological tests due to a language barrier or a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).
11. Cognitive impairment or physical impairment such that they are unable to learn to, or physically unable to apply tDCS to their scalp without assistance (after training).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients maintaining remission of depressive symptoms or response to rTMS treatments as measured by the Hamilton Rating Scale for Depression - 17 Hamilton Rating Scale for Depression (17-item version) | 6 months
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-52 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)

SECONDARY OUTCOMES:
Proportion of responders and remitters who relapse | 6 months
  Relapse defined separately for responders and remitters Responders who experience >50% worsening of their HRSD-17 scores from baseline, over 2 consecutive assessments, will discontinue tDCS and discuss treatment options with a study physician. Remitters will discontinue tDCS and discuss treatment options if they have an HRSD-17 score of >18 over 2 consecutive assessments separated by at least 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research